CLINICAL TRIAL: NCT02486640
Title: BETAPREDICT - MS Patients Treated With BETAferon®: PREDICTors of Treatment Adherence
Brief Title: Evaluation of Potential Predictors of Adherence by Investigating a Representative Cohort of Multiple Sclerosis (MS) Patients in Germany Treated With Betaferon
Acronym: BETAPREDICT
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18016; BF1502 (Registry Identifier: NIS Trial Alias)
Record Dates: First submitted 2015-06-15; First posted 2015-07-01 (Estimated); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Multiple Sclerosis
Keywords: RRMS, CIS
MeSH Terms: conditions — Multiple Sclerosis; Carcinoma in Situ | interventions — Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Betaferon
  Interventions: Drug: Interferon beta-1b (Betaferon, BAY86-5046); Device: Betaconnect Autoinjector

INTERVENTIONS:
Drug: Interferon beta-1b (Betaferon, BAY86-5046) — Multiple Sclerosis patients who are treated with Betaferon and who are using the Betaconnect autoinjector.
Device: Betaconnect Autoinjector — Multiple Sclerosis patients who are treated with Betaferon and who are using the Betaconnect autoinjector.

SUMMARY:
This study aims to evaluate potential predictors of adherence by investigating a representative cohort of MS patients in Germany treated with Betaferon

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years with the diagnosis of relapsing remitting multiple sclerosis or a clinically isolated syndrome
* Patients on treatment with Betaferon or the decision to treat patients with Betaferon has been made by the attending physician
* Patients using or willing to use the BETACONNECT autoinjector for Betaferon application
* Written informed consent

Exclusion Criteria:

* Patients receiving any other disease modifying drug
* Contraindications of Betaferon described in the Summary of Product Characteristics
* Patients participating in any other clinical or non-interventional study, evaluating MS therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients with relapsing remitting multiple sclerosis (RRMS) or patients with a clinically isolated syndrome (CIS) who are treated with Betaferon or will be treated with Betaferon according to the attending physician's decision and for whom the patient and the physician have agreed to use the BETACONNECT device
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2015-09-08 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
Compliance to therapy (%) | 12 months
  Compliance (%) = ((expected # of treatment days during observation period - missed # of treatment days during observation period)/(expected # of treatment days during observation period))*100
Persistence of therapy (Yes or No) | 12 months
  Persistence is defined as patients continuing ("persisting") their medication (regardless of the frequency of intake)
Overall adherence to therapy (Yes or No) | 12 months
  Patients will be defined as being adherent to therapy if they fulfill the following criteria: a. They have been at least 80% compliant, i.e. injected ≥80% of the expected Betaferon dosages and b. They have not dropped out of the study prior to the time of evaluation (i.e. they did not stop Betaferon treatment for any reason including switching to another medication prior to the time of evaluation).

SECONDARY OUTCOMES:
Satisfaction with the BETACONNECT autoinjector, recorded by the patient questionnaire | Up to 24 months
Adherence to Betaferon treatment is associated with: depression, health related quality of life, coping mechanisms, self-management mechanisms, social support, fatigue, and cognition. (Yes or No) | Up to 24 months
Adherence to Betaferon treatment is associated with number of relapses (Yes or No) | 12 months, 24 months
Adherence to Betaferon treatment is associated with EDSS change (Yes or No) | 12 months, 24 months
  EDSS (Expanded Disability Status Scale)
Adherence to Betaferon treatment is associated with utilities of treatment, recorded by the EQ-5D quality of life questionnaire (Yes or No) | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Wermsdorf, Saxony, Germany

REFERENCES:
- [Derived] Kohler W, Bayer-Gersmann K, Neusser T, Schurks M, Ziemssen T. Predictors of Adherence Among Patients With Multiple Sclerosis Using the BETACONNECT(R) Autoinjector: A Prospective Observational Cohort Study. Front Neurol. 2021 Feb 24;12:643126. doi: 10.3389/fneur.2021.643126. eCollection 2021. PMID 33716945